CLINICAL TRIAL: NCT00313716
Title: Effects of Erythropoietin on Cerebral Vascular Dysfunction and Anemia in Traumatic Brain Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Claudia Sue Robertson (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Claudia Sue Robertson, Professor, Department of Neurosurgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: P01NS038660 (NIH); P01NS038660 (NIH)
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Anemia; Traumatic Brain Injury
Keywords: anemia; traumatic brain injury; recombinant human erythropoietin; rhEpo; erythropoietin; TBI; Epo
MeSH Terms: conditions — Anemia; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Epo1 and TT10 (Active Comparator): recombinant human erythropoietin, rhEpo administration (500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury) and hemoglobin transfusion trigger of 10gm/dl
  Interventions: Drug: recombinant human erythropoietin, rhEpo
- Epo1 and TT7 (Active Comparator): recombinant human erythropoietin, rhEpo administration (500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury) and hemoglobin transfusion trigger 7gm/dl
  Interventions: Drug: recombinant human erythropoietin, rhEpo
- Epo2 and TT10 (Active Comparator): recombinant human erythropoietin, rhEpo administration (500 IU/kg within 6 hrs of injury, and at 9 and 16 days after injury) and hemoglobin transfusion trigger 10gm/dl
  Interventions: Drug: recombinant human erythropoietin, rhEpo
- Epo2 and TT7 (Active Comparator): recombinant human erythropoietin, rhEpo administration (500 IU/kg within 6 hrs of injury, and at 9 and 16 days after injury) and hemoglobin transfusion trigger 7gm/dl
  Interventions: Drug: recombinant human erythropoietin, rhEpo
- Placebo and TT10 (Placebo Comparator): Placebo administration and transfusion threshold 10 gm/dl
  Interventions: Other: placebo
- Placebo and TT7 (Placebo Comparator): Placebo administration and transfusion threshold 7 gm/dl
  Interventions: Other: placebo

INTERVENTIONS:
Drug: recombinant human erythropoietin, rhEpo — The study design is 2x2 factorial with randomization to erythropoietin or placebo and to transfusion trigger 10 gm/dl or 7 g/dl. Erythropoietin or placebo was initially dosed daily for 3 days and then weekly for 2 more weeks (first 74 patients, Epo1 dosing regimen), and then the 24- and 48-hour doses were stopped for the remainder of the patients (remaining 126 patients, Epo2 dosing regimen).
  Arms: Epo1 and TT10; Epo1 and TT7; Epo2 and TT10; Epo2 and TT7
Other: placebo — an inactive substance
  Arms: Placebo and TT10; Placebo and TT7

SUMMARY:
The purpose of this study is to determine the effect of early administration of recombinant human erythropoietin on long-term neurological outcome after severe traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) causes a spectrum of cerebrovascular dysfunction, ranging from impaired pressure autoregulation to severe global ischemia (inadequate blood flow). Pressure autoregulation is the ability of an organ to maintain a constant blood flow despite changes in perfusion pressure. Impaired pressure autoregulation causes TBI patients to be more vulnerable to secondary ischemic attacks.

Erythropoietin (Epo) is a substance that is normally made by the kidneys and stimulates the production of red blood cells. It is usually given to patients to treat anemia. Scientists recently discovered that Epo also is made in the brain after injury. In animal models of TBI, the brain's production of Epo has numerous protective effects, including reducing inflammation in the brain, reducing death of brain cells, and improving blood flow to the brain. In the laboratory, the effects of this naturally-occurring, protective agent can be enhanced by giving additional amounts intravenously. Because Epo may have beneficial effects for both the injured brain and anemia, scientists are studying the effects of giving Epo to patients with severe TBI.

The primary objective of this randomized, placebo-controlled study is to determine the effect of early administration of recombinant human Epo (rhEpo), on long-term neurological outcome in patients with severe TBI. The researchers also will examine the effects of rhEpo administration on the cerebrovascular system, hemoglobin concentration, brain oxygenation, the need for blood transfusion, and on systemic complications.

This study consists of 2 parts: 1) a treatment phase, and 2) a monitoring phase. In the treatment phase, participants will be randomly assigned to 1 of 4 groups: a low or high dose rhEPO treatment group or low or high dose placebo group (control group). All other aspects of treatment during the acute post-injury phase will follow the standard treatment protocol for individuals with severe TBI. Generally the treatment phase lasts 1-2 weeks or the amount of time that is required for patients to receive treatment of their TBIs in the ICU (intensive care unit). The monitoring part of the study (which includes recording information from tests performed as part of the standard TBI treatment, as well as some additional tests performed especially for the study) lasts for up to 6 months after the TBI.

Information learned in this study may lead to knowledge about whether rhEpo improves outcomes after TBI and about the optimal hemoglobin concentration to maintain in patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

* Blunt trauma mechanism of brain injury
* Glasgow Coma Score - motor component ≤ 5 (not following commands) on the post-resuscitation neurologic exam
* Available for enrollment and administration of study drug within 6 hours of injury

Exclusion Criteria:

* Penetrating trauma (i.e. gun shot wounds)
* Glasgow Coma Score = 3 and bilateral fixed and dilated pupils
* Abbreviated Injury Scale score > 5 for any body part except brain
* Severe pre-existing chronic disease
* Uncontrolled hypertension, defined as mean arterial pressure > 130mmHg despite antihypertensive treatment
* Known hypersensitivity to mammalian cell-derived products or human albumin
* Currently taking anticoagulants

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Robertson, MD, Principal Investigator — Professor, Department of Neurosurgery, Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Ben Taub General Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Robertson CS, Hannay HJ, Yamal JM, Gopinath S, Goodman JC, Tilley BC; Epo Severe TBI Trial Investigators; Baldwin A, Rivera Lara L, Saucedo-Crespo H, Ahmed O, Sadasivan S, Ponce L, Cruz-Navarro J, Shahin H, Aisiku IP, Doshi P, Valadka A, Neipert L, Waguspack JM, Rubin ML, Benoit JS, Swank P. Effect of erythropoietin and transfusion threshold on neurological recovery after traumatic brain injury: a randomized clinical trial. JAMA. 2014 Jul 2;312(1):36-47. doi: 10.1001/jama.2014.6490. PMID 25058216
- [Derived] Aisiku IP, Yamal JM, Doshi P, Benoit JS, Gopinath S, Goodman JC, Robertson CS. Plasma cytokines IL-6, IL-8, and IL-10 are associated with the development of acute respiratory distress syndrome in patients with severe traumatic brain injury. Crit Care. 2016 Sep 15;20:288. doi: 10.1186/s13054-016-1470-7. PMID 27630085
- [Derived] Yamal JM, Benoit JS, Doshi P, Rubin ML, Tilley BC, Hannay HJ, Robertson CS. Association of transfusion red blood cell storage age and blood oxygenation, long-term neurologic outcome, and mortality in traumatic brain injury. J Trauma Acute Care Surg. 2015 Nov;79(5):843-9. doi: 10.1097/TA.0000000000000834. PMID 26496111
- [Derived] Aisiku IP, Yamal JM, Doshi P, Rubin ML, Benoit JS, Hannay J, Tilley BC, Gopinath S, Robertson CS. The incidence of ARDS and associated mortality in severe TBI using the Berlin definition. J Trauma Acute Care Surg. 2016 Feb;80(2):308-12. doi: 10.1097/TA.0000000000000903. PMID 26491799
- [Derived] Yamal JM, Robertson CS, Rubin ML, Benoit JS, Hannay HJ, Tilley BC. Enrollment of racially/ethnically diverse participants in traumatic brain injury trials: effect of availability of exception from informed consent. Clin Trials. 2014 Apr;11(2):187-94. doi: 10.1177/1740774514522560. PMID 24686108

RESULTS

PARTICIPANT FLOW:
Groups:
- Epo1/TT7 Arm: High dose Epo (patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury) and hemoglobin transfusion threshold 7 gm/dl
- Epo2/TT7 Arm: Low dose Epo (patients received erythropoietin 500 IU/kg within 6 hrs of injury, and at 9 and 16 days after injury) and hemoglobin transfusion threshold 7 gm/dl
- Placebo/TT7 Arm: Placebo (patients received saline) and hemoglobin transfusion threshold 7 gm/dl
- Epo1/TT10 Arm: High dose Epo (patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury) and hemoglobin transfusion threshold 10 gm/dl
- Epo2/TT10 Arm: Low dose Epo (patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury) and hemoglobin transfusion threshold 10 gm/dl
- Placebo/TT10 Arm: Placebo (patients received saline) and hemoglobin transfusion threshold 10 gm/dl
Period: Overall Study
Arm/Group | Epo1/TT7 Arm | Epo2/TT7 Arm | Placebo/TT7 Arm | Epo1/TT10 Arm | Epo2/TT10 Arm | Placebo/TT10 Arm
Started | 18 | 31 | 50 | 20 | 33 | 48
Completed | 13 | 23 | 38 | 16 | 27 | 35
Not Completed | 5 | 8 | 12 | 4 | 6 | 13
Not completed — Death | 3 | 2 | 9 | 3 | 5 | 9
Not completed — Lost to Follow-up | 2 | 5 | 2 | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Epo1/TT7 Arm: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury and transfused to keep hemoglobin at least 7 g/dl
- Epo2/TT7 Arm: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury and transfused to keep hemoglobin concentration at least 7 g/dl
- Placebo/TT7 Arm: Patients received saline and transfused to keep hemoglobin concentration at least 7 g/dl
- Epo1/TT10 Arm: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury and transfused to keep hemoglobin at least 10 g/dl
- Epo2/TT10 Arm: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury and transfused to keep hemoglobin concentration at least 10 g/dl
- Placebo/TT10 Arm: Patients received saline and transfused to keep hemoglobin concentration at least 10 g/dl
- Total: Total of all reporting groups
Arm/Group | Epo1/TT7 Arm | Epo2/TT7 Arm | Placebo/TT7 Arm | Epo1/TT10 Arm | Epo2/TT10 Arm | Placebo/TT10 Arm | Total
Number analyzed (Participants) | 18 | 31 | 50 | 20 | 33 | 48 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.5 [22 to 52] | 28 [23 to 48] | 29.5 [20 to 39] | 36.5 [28.5 to 44] | 30 [23 to 46] | 30.5 [25 to 45] | 30 [23 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 9 | 2 | 5 | 5 | 26
  Male | 16 | 28 | 41 | 18 | 28 | 43 | 174
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 1 | 0 | 0 | 3 | 6
  Hispanic | 8 | 16 | 26 | 12 | 19 | 22 | 103
  Black | 4 | 4 | 12 | 3 | 6 | 14 | 43
  White, non-Hispanic | 5 | 10 | 11 | 5 | 8 | 9 | 48
Prehospital hypotension [Number; unit: participants]
  yes | 1 | 3 | 7 | 3 | 2 | 9 | 25
  no | 17 | 28 | 43 | 17 | 31 | 39 | 175
Prehospital hypoxia [Number; unit: participants]
  yes | 0 | 2 | 16 | 3 | 5 | 13 | 39
  no | 18 | 29 | 34 | 17 | 28 | 35 | 161
Mechanism of injury [Number; unit: participants]
  Assault | 0 | 2 | 5 | 2 | 3 | 10 | 22
  Fall or jump | 8 | 3 | 7 | 3 | 4 | 2 | 27
  Automobile crash | 10 | 19 | 29 | 9 | 22 | 27 | 116
  Motorcycle crash | 0 | 7 | 7 | 5 | 4 | 8 | 31
  Other | 0 | 0 | 2 | 1 | 0 | 1 | 4
Injury Severity Score [Median (Inter-Quartile Range); unit: units on a scale] — Injury Severity Score describes the severity of all traumatic injuries. The score ranges from 0 to 75, with a higher score indicating a more severe injury.
  units on a scale | 29 [26 to 34] | 30 [25 to 35] | 29 [25 to 43] | 27 [26 to 36.5] | 29 [25 to 38] | 29 [25 to 35] | 29 [25 to 36.5]
IMPACT probability of poor outcome [Mean (Standard Deviation); unit: probability of poor outcome] | .29 (.2) | .35 (.2) | .45 (.3) | .49 (.2) | .46 (.3) | .38 (.3) | .41 (.25)
Motor component of Glasgow Coma Score [Number; unit: participants] — The motor component of the Glasgow Coma Score describes the motor response. The scale ranges from 1-6 (1=no response, 2=decerebrate posturing, 3=decorticate posturing, 4=withdrawal response, 5=localizing response, 6=following commands) with a higher score indicating better performance.
  participants
    mGCS 1-3 | 4 | 12 | 20 | 8 | 14 | 13 | 71
    mGCS 4-5 | 14 | 19 | 30 | 12 | 19 | 35 | 129
Sum Glasgow Coma Score [Number; unit: participants] — The Sum Glasgow Coma Score sums the three components of the neurological examination (eye, verbal, and motor responses). The score ranges from 3 to 15 with 3 indicating no response, and 15 indicating normal response.
  participants
    GCS 3-5 | 4 | 10 | 20 | 8 | 13 | 11 | 66
    GCS 6-8 | 10 | 13 | 19 | 8 | 16 | 23 | 89
    GCS > 8 | 4 | 8 | 11 | 4 | 4 | 14 | 45
Pupil reactivity [Number; unit: participants]
  Both reactive | 12 | 24 | 27 | 13 | 17 | 28 | 121
  One reactive | 2 | 4 | 8 | 3 | 1 | 5 | 23
  Neither reactive | 4 | 3 | 15 | 4 | 15 | 15 | 56
Marshall CT scan category [Number; unit: participants] — Marshall CT scan category is a classification system for traumatic brain injury. Diffuse injury 1 is a normal scan. Diffuse injury 2 has some abnormalities but basal cisterns are present. Diffuse injury 3 has basal cistern compression but no midline shift. Diffuse injury 4 has midline shift. Mass lesions include hematomas and contusions of at least 25 ml in volume.
  participants
    Diffuse injury 1 or 2 | 10 | 15 | 24 | 5 | 15 | 20 | 89
    Diffuse injury 3 or 4 | 5 | 8 | 10 | 9 | 2 | 12 | 46
    Mass lesion | 3 | 8 | 16 | 6 | 16 | 16 | 65
Presence of subarachnoid hemorrhage [Number; unit: participants]
  yes | 12 | 22 | 37 | 3 | 22 | 11 | 107
  no | 6 | 9 | 13 | 17 | 11 | 37 | 93
Presence of epidural hematoma [Number; unit: participants]
  yes | 3 | 4 | 3 | 3 | 8 | 11 | 32
  no | 15 | 27 | 47 | 17 | 25 | 37 | 168
Hemoglobin concentration [Median (Inter-Quartile Range); unit: g/dl] | 14.7 [13.9 to 16.0] | 14.7 [13.2 to 15.5] | 14.0 [12.3 to 15.6] | 14.8 [13.0 to 15.6] | 13.9 [12.7 to 15.4] | 14.7 [13.6 to 15.6] | 14.45 [12.95 to 15.6]
Glucose concentration [Median (Inter-Quartile Range); unit: mmol/L] | 8.3 [7.2 to 10.2] | 9.1 [7.2 to 10.6] | 8.9 [7.5 to 10.4] | 8.8 [7.4 to 11.7] | 8.6 [7.1 to 9.7] | 7.7 [6.6 to 10.0] | 8.42 [7.11 to 10.22]
Surgery on admission [Number; unit: participants]
  Evacuation epidural hematoma | 0 | 2 | 1 | 0 | 1 | 5 | 9
  Evacuation subdural hematoma | 2 | 5 | 13 | 5 | 14 | 7 | 46
  Evacuation intracerebral hematoma or contusion | 1 | 0 | 1 | 1 | 0 | 1 | 4
  Non-central nervous system injury | 0 | 0 | 1 | 0 | 0 | 1 | 2
  No surgery on admission | 15 | 24 | 34 | 14 | 18 | 34 | 139

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale
Description: Dichotomized to favorable outcome (good recovery or moderate disability) or to unfavorable outcome (severe disability or vegetative or dead)
Time Frame: at 6 months after injury
Population: Intention to treat. Multiple imputation for missing 6-month GOS data was performed assuming data were missing at random using chained equations (R, R Foundation for Statistical Computing).The imputation was based on a logistic regression model with baseline covariates. Results were aggregated over 20 imputed sets using variance formula by Rubin.
Measure: Number; unit: participants
Groups:
- Epo1 Group: Patients received erythropoietin 500 IU/kg within 6hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury (Epo1/TT10 arm and Epo1/TT7 arm combined)
- Epo2 Group: Patients received erythropoietin 500 IU/kg within 6hrs of injury, and at 9 and 16 days after injury (Epo2/TT10 arm and Epo2/TT7 arm combined)
- Placebo Group: Patients received saline (Placebo/TT10 arm and Placebo/TT7 arm combined)
- TT7 Group: Patients had hemoglobin concentration maintained at least 7 gm/dl (Epo1/TT7 arm, Epo2/TT7 arm, and Placebo/TT7 arm combined)
- TT10 Group: Patients had hemoglobin concentration maintained at least 10 gm/dl (Epo1/TT10 arm, Epo2/TT10 arm, and Placebo/TT10 arm combined)
Arm/Group | Epo1 Group | Epo2 Group | Placebo Group | TT7 Group | TT10 Group
Number analyzed (Participants) | 35 | 57 | 89 | 87 | 94
participants
  Favorable outcome | 17 | 17 | 34 | 37 | 31
  Unfavorable outcome | 18 | 40 | 55 | 50 | 63
Statistical Analysis 1: Comparison: Epo2 Group vs Placebo Group; The primary analysis plan was a futility trial of the Epo 2 regimen arm. We hypothesized that 30% of subjects in the placebo group would have a favorable outcome at six months and there would be no interaction between the Epo and the transfusion threshold groups. Using a one-sided alpha of 0.15, a sample size of 62 subjects in the Epo 2 regimen group and 100 subjects in the placebo group provided 91% power to test the futility hypothesis; Test type: Superiority or Other; p = .01, Futility analysis — H0: Proportion of participants expected to have a favorable GOS outcome in the Epo2 group - in Placebo group is >= 0.2. H1: Proportion in Epo2 group - in Placebo group < 0.2
Statistical Analysis 2: Comparison: Epo1 Group vs Placebo Group; The primary analysis plan was a futility trial of the Epo 1 regimen arm. We hypothesized that 30% of subjects in the placebo group would have a favorable outcome at six months and there would be no interaction between the Epo and the transfusion threshold groups; Test type: Superiority or Other; p = 0.13, Futility analysis — H0: Proportion of participants expected to have a favorable GOS outcome in the Epo1 group - in Placebo group is >= 0.2. H1: Proportion in Epo1 group - in Placebo group < 0.2
Statistical Analysis 3: Comparison: TT7 Group vs TT10 Group; We hypothesized that 40% of the patients in the TT7 group would have a favorable GOS score and that there would be no interaction between the Epo and TT groups. Assuming a 2-sided test with an alpha level of 0.05, we estimated that a sample size of 200 patients would provide 80% power to detect a 20% absolute increase in the GOS score for the TT10 group; Test type: Superiority or Other; p = .34, 2-sample test of proportions

2. Secondary Outcome: Disability Rating Scale
Description: Disability rating scale was a secondary outcome measure for the transfusion threshold analysis. Disability rating scale ranges from 0 to 30, with 30 indicating death and 0 indicating return to normal status.
Time Frame: at 6 months
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TT7 Group | TT10 Group
Number analyzed (Participants) | 87 | 94
units on a scale | 5 [2.25 to 9.75] | 8 [4 to 17]
Statistical Analysis 1: Comparison: TT7 Group vs TT10 Group; Test type: Superiority or Other; p = .06, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mortality Rate
Description: mortality rate was a secondary outcome measure for the Epo randomization, and a primary safety outcome measure for the transfusion threshold randomization
Time Frame: up to 6 months after injury
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- Epo1 Group: Patients received 500 IU/kg erythropoietin within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury (Epo1/TT10 arm and Epo1/TT7 arm combined)
- Epo2 Group: Patients received 500 IU/kg within 6 hrs after injury, and at 9 and 16 days after injury (Epo2/TT10 arm and Epo2/TT7 arm combined)
- TT7 Group: Patients had hemoglobin maintained at least 7 gm/dl (Epo1/TT7 arm, Epo2/TT7 arm, and Placebo/TT7 arm combined)
Arm/Group | Epo1 Group | Epo2 Group | Placebo Group | TT7 Group | TT10 Group
Number analyzed (Participants) | 38 | 64 | 98 | 99 | 101
participants
  Died | 6 | 7 | 18 | 14 | 17
  Survived | 32 | 57 | 80 | 85 | 84
Statistical Analysis 1: Comparison: Epo2 Group vs Placebo Group; Test type: Superiority or Other; p = .25, Log Rank
Statistical Analysis 2: Comparison: Epo1 Group vs Placebo Group; Test type: Superiority or Other; p = .75, Log Rank
Statistical Analysis 3: Comparison: TT7 Group vs TT10 Group; Test type: Superiority or Other; p = .72, Log Rank

4. Secondary Outcome: Incidence of Adult Respiratory Distress Syndrome (ARDS)
Description: development of ARDS was a primary safety outcome for the transfusion threshold randomization
Time Frame: within 30 days after injury
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | TT7 Group | TT10 Group
Number analyzed (Participants) | 99 | 101
participants
  Developed ARDS | 16 | 25
  Did not develop ARDS | 83 | 76
Statistical Analysis 1: Comparison: TT7 Group vs TT10 Group; Test type: Superiority or Other; p = .08, Regression, Cox; Hazard Ratio (HR) = 1.79, 95% CI 2-sided [.93 to 3.45]

5. Secondary Outcome: Incidence of Infection
Description: occurrence of infection was a primary safety outcome for the transfusion threshold randomization
Time Frame: within 30 days after injury
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- TT10 Group: Patients had hemoglobin concentration maintained at least 10 gm/dl (Epo1/TT10 group, Epo2/TT10 group, and Placebo/TT10 group combined)
Arm/Group | TT7 Group | TT10 Group
Number analyzed (Participants) | 99 | 101
participants
  Developed one or more infections | 27 | 36
  Did not develop infection | 72 | 65
Statistical Analysis 1: Comparison: TT7 Group vs TT10 Group; Test type: Superiority or Other; p = .26, 2-sample test - equality of proportions; Mean Difference (Final Values) = -.08, 95% CI 2-sided [-.22 to .05]

ADVERSE EVENTS:
Time Frame: Serious adverse events were reported for 30 days after injury
Description: Each patient is represented twice in the table (once in the Epo1/Epo2/Placebo groups and once in the TT7/TT10 groups)
Groups:
- Epo1 Group: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, at 24 and 48 hrs after injury, and at 9 and 16 days after injury (Epo1/TT10 arm and Epo1/TT7 arm combined)
- Epo2 Group: Patients received erythropoietin 500 IU/kg within 6 hrs of injury, and at 9 and 16 days after injury (Epo1/TT10 arm and Epo1/TT7 arm combined)
Arm/Group | Epo1 Group | Epo2 Group | Placebo Group | TT7 Group | TT10 Group
Serious Adverse Events (participants affected / at risk) | 29/38 | 50/64 | 78/98 | 85/99 | 93/101
Other Adverse Events (participants affected / at risk) | 34/38 | 57/64 | 87/98 | 85/99 | 93/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epo1 Group (N=38) | Epo2 Group (N=64) | Placebo Group (N=98) | TT7 Group (N=99) | TT10 Group (N=101)
Brain death (Nervous system disorders) | 3 | 2 | 5 | 6 | 4
Brain tissue hypoxia (Nervous system disorders) | 3 | 4 | 8 | 10 | 5 — Brain tissue pO2 less than 10 mmHg for more than 10 minutes
delayed or recurrent intracranial hemorrhage (Nervous system disorders) | 10 | 13 | 18 | 15 | 26 — new hematoma or increase in hematoma after initial CT scan, or recurrence of a hematoma after surgical evacuation
hydrocephalus (Nervous system disorders) | 1 | 2 | 2 | 3 | 2
intracranial hypertension (Nervous system disorders) | 7 | 14 | 28 | 22 | 27 — intracranial hypertension requiring treatment with mannitol, barbiturate coma, decompressive craniectomy or that resulted in neurological deterioration or death
meningitis or ventriculitis (Nervous system disorders) | 2 | 2 | 2 | 3 | 3
wound dehiscence (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
stroke (Nervous system disorders) | 3 | 0 | 0 | 1 | 2
Lower extremity deep venous thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 1 | 1
cardiac arrest with CPR (Cardiac disorders) | 2 | 1 | 2 | 2 | 3
Gangrene of extremities (Vascular disorders) | 2 | 0 | 0 | 0 | 2
Hypotension due to barbiturate coma (Cardiac disorders) | 2 | 4 | 6 | 3 | 9
Upper extremity deep venous thrombophlebitis (Vascular disorders) | 1 | 1 | 0 | 0 | 2
Pulmonary embolus (Cardiac disorders) | 0 | 4 | 3 | 1 | 6
Shock (Cardiac disorders) | 10 | 15 | 19 | 25 | 19 — Hypotension (mean blood pressure less than 60 mmHg) requiring treatment with pressors
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3
peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Severe anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 — Hemoglobin concentration less than 6 gm/dl
Other severe hematologic disorder (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3 | 3
Multiple organ dysfunction syndrome (Infections and infestations) | 0 | 1 | 2 | 0 | 3
Wound infection, non-central nervous system (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 11 | 8 | 14 | 13 | 20
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 2 | 1 | 3 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 2 | 8 | 7 | 4
Carotid cavernous fistula (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Infected eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Hemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Osteomyelitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Rhabdomyalysis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Tongue laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
internal jugular vein injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Acute renal failure (Renal and urinary disorders) | 2 | 1 | 3 | 3 | 3
Severe metabolic acidosis (Renal and urinary disorders) | 1 | 0 | 2 | 1 | 2
Severe mixed acid-base disorder (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 2 | 9
Airway obstruction post-extubation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 1
Severe atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1
Electrolyte disturbance (Renal and urinary disorders) | 0 | 4 | 7 | 5 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epo1 Group (N=38) | Epo2 Group (N=64) | Placebo Group (N=98) | TT7 Group (N=99) | TT10 Group (N=101)
Cerebrospinal fluid leak (Nervous system disorders) | 2 | 1 | 2 | 1 | 4
Brain tissue hypoxia (Nervous system disorders) | 9 | 12 | 21 | 21 | 21
Delayed or recurrent intracranial hematoma (Nervous system disorders) | 7 | 5 | 12 | 11 | 13
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Intracranial hypertension (Nervous system disorders) | 9 | 9 | 15 | 17 | 16
Pneumocephalus (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1
Seizure (Nervous system disorders) | 3 | 3 | 5 | 4 | 7
Subgaleal cerebrospinal fluid collection (Nervous system disorders) | 1 | 0 | 1 | 1 | 1
Lower extremity deep venous thrombophlebitis (Vascular disorders) | 1 | 2 | 4 | 2 | 5
Atrial arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Cardiac disorders) | 1 | 1 | 0 | 0 | 2
Hypotension from barbiturate coma (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Upper extremity deep vein thrombophlebitis (Vascular disorders) | 7 | 7 | 6 | 10 | 10
Hypotension (Cardiac disorders) | 1 | 0 | 2 | 3 | 0
Upper GI bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Elevated transaminases (Hepatobiliary disorders) | 11 | 14 | 26 | 25 | 26
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 24 | 33 | 60 | 66 | 51
Other hematologic disorder (Blood and lymphatic system disorders) | 13 | 20 | 43 | 37 | 39
Urinary tract infection (Infections and infestations) | 1 | 5 | 7 | 7 | 6
Bacteremia (Infections and infestations) | 0 | 1 | 3 | 2 | 2
Wound infection, non-central nervous system (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1 | 1 | 0
Diffuse edema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyperglycemia (Endocrine disorders) | 3 | 0 | 4 | 4 | 3
Hypoglycemia (Endocrine disorders) | 0 | 1 | 2 | 1 | 2
Hypothermia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1
Bleeding complicating a procedure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 2
Exposure keratoconjunctivitis (Eye disorders) | 1 | 0 | 2 | 2 | 1
Rhabdomyalysis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
acute renal dysfunction (Renal and urinary disorders) | 0 | 0 | 5 | 4 | 1
Metabolic acidosis (Renal and urinary disorders) | 3 | 0 | 4 | 4 | 3
Mixed acid-base abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Airway obstruction post-extubation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 14 | 14 | 19 | 21 | 26
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6 | 4 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 6 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 3
Febrile transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Electrolyte imbalance (Renal and urinary disorders) | 12 | 20 | 36 | 28 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No